CLINICAL TRIAL: NCT03183115
Title: Preemptive Radiofrequency Ablation for Esophageal Speckled Lugol Background Mucosa to Prevent Metachronous Neoplastic Recurrence After Complete Endoscopic Submucosal Dissection ~A Randomized Controlled Study
Brief Title: RFA to Prevent Metachronous Squamous Neoplasia Recurrence After Complete Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ED102807; MOST105-2314-B-650-005 (Other Grant/Funding Number: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2017-05-28; First posted 2017-06-09 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Squamous Cell Neoplasm
Keywords: Early esophageal squamous cell neoplasm; Radiofrequency ablation; Endoscopic submucosal dissection; Esophageal cancer; Recurrence; Field cancerization
MeSH Terms: conditions — Esophageal Neoplasms; Recurrence | interventions — Radiofrequency Ablation; Endoscopy; Lugol's solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA group (Experimental): Balloon type RFA (12J/cm2, 1 application) will be applied for the entire speckled esophageal mucosa at the 3 months after complete ESD.
  Oral prednisolone 30mg/day will be prescribed at day 3 after RFA procedure and continue for 28 days to prevent the post-RFA stenosis.
  Interventions: Procedure: Radiofrequency ablation; Device: Endoscopy; Drug: Lugol's Solution (1.5%)
- Control group (No Intervention): No intervention; surveillance endoscopy alone

INTERVENTIONS:
Procedure: Radiofrequency ablation — HALO360 System (Covidien GI Solutions, Sunnyvale, California, USA), which has been approved by the US Food and Drug Administration (FDA) and is approved for use in Europe (CE mark) and Taiwan (Ministry of Health and Welfare). Because the HALO 360 balloon catheter has been phased out since 2019, a new Barrx™ 360 Express catheter was used thereafter.
  Arms: RFA group
Device: Endoscopy — The participants will receive meticulous endoscopic examination with Lugol chromoendoscopy and Narrow-band imaging
  Arms: RFA group
Drug: Lugol's Solution (1.5%) — Before the RFA intervention, the participants will received Lugol staining over the esophagus
  Arms: RFA group

SUMMARY:
Esophageal cancer is a highly lethal disease, and its incidence is still increasing in the world. Recent advances in image-enhanced techniques such as Lugol chromoendoscopy and narrow band imaging, the number of patients with early esophageal squamous cell neoplasias (ESCNs) detected has markedly increased. Endoscopic submucosal dissection (ESD) enables en bloc resection of the neoplasia, and the resected specimen allows for a pathological assessment to evaluate the curability. However, the patients who received complete ESD for early ESCNs frequently developed metachronous recurrence. The cumulative metachronous recurrence rate at 5 years was 50%, and the mean annual incidence of newly diagnosed metachronous tumors was 10%. Among them, those with "speckled" lugol staining pattern over the esophageal background mucosa have the highest risk and should be seen as a precancerous lesion of ESCCs. This issue is gaining attention in the era of endoscopic treatment, but currently there was no appropriate strategy to prevent the tumor recurrence in these high-risk subjects.

Endoscopic radiofrequency ablation (RFA) is a rapidly evolving therapeutic modality, and recent studies have shown its efficacy and safety for eradicating for flat type early ESCNs. To search a best strategy for the prevention of ESCNs, the investigators thus propose a hypothesis that the preemptive RFA for esophageal "speckled" lugol background mucosa may prevent the metachronous neoplastic recurrence after complete endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

* Adults with early stage ESCNs (squamous high grade dysplasia, carcinoma in situ, or T1N0M0 SCC) who were treated by endoscopic submucosal dissection.
* Lugol staining showed "speckled" (>10 small lugol-unstained lesions) pattern of background mucosa.

Exclusion Criteria:

* Having a history of incomplete endoscopic treatment, or complications during/after treatment (perforation, stricture).
* Having history of systemic chemotherapy or radiation therapy for esophagus or post esophagectomy.
* Life expectancy <2 yr.
* Decompensated cirrhosis (Child score B, C).
* Having large esophageal varices.
* Poor performance status (ECOG>2).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence | From date of randomization until the date of first documented tumor recurrence, assessed up to 100 months
  Metachronous tumor recurrence is defined as a tumor (high-grade dysplasia or squamous cell carcinoma) recurring at a new site after more than 6 months of complete remission status.

SECONDARY OUTCOMES:
Major adverse events | From date of intervention until the date of first documented adverse events, assessed up to 12months
  including perforation, dysphagia, stenosis, defined as the failure of a standard endoscope (9.8 mm in diameter) to pass through the stenosis, or others resulting in the patients intolerable and discontinued intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- EDA Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The initial outcome and the data of adverse events will be shared with other researchers, by mail, when they are available.

REFERENCES:
- [Result] Lee CT, Chang CY, Lee YC, Tai CM, Wang WL, Tseng PH, Hwang JC, Hwang TZ, Wang CC, Lin JT. Narrow-band imaging with magnifying endoscopy for the screening of esophageal cancer in patients with primary head and neck cancers. Endoscopy. 2010 Aug;42(8):613-9. doi: 10.1055/s-0030-1255514. Epub 2010 Jul 28. PMID 20669074
- [Result] Lee CT, Chang CY, Tai CM, Wang WL, Tseng CH, Hwang JC, Lin JT. Endoscopic submucosal dissection for early esophageal neoplasia: a single center experience in South Taiwan. J Formos Med Assoc. 2012 Mar;111(3):132-9. doi: 10.1016/j.jfma.2010.12.002. Epub 2012 Feb 8. PMID 22423666
- [Result] Shimizu Y, Tukagoshi H, Fujita M, Hosokawa M, Kato M, Asaka M. Metachronous squamous cell carcinoma of the esophagus arising after endoscopic mucosal resection. Gastrointest Endosc. 2001 Aug;54(2):190-4. doi: 10.1067/mge.2001.116877. PMID 11474389
- [Result] Urabe Y, Hiyama T, Tanaka S, Oka S, Yoshihara M, Arihiro K, Chayama K. Metachronous multiple esophageal squamous cell carcinomas and Lugol-voiding lesions after endoscopic mucosal resection. Endoscopy. 2009 Apr;41(4):304-9. doi: 10.1055/s-0029-1214477. Epub 2009 Apr 1. PMID 19340732
- [Result] Muto M, Hironaka S, Nakane M, Boku N, Ohtsu A, Yoshida S. Association of multiple Lugol-voiding lesions with synchronous and metachronous esophageal squamous cell carcinoma in patients with head and neck cancer. Gastrointest Endosc. 2002 Oct;56(4):517-21. doi: 10.1067/mge.2002.128104. PMID 12297767
- [Result] Shaheen NJ, Sharma P, Overholt BF, Wolfsen HC, Sampliner RE, Wang KK, Galanko JA, Bronner MP, Goldblum JR, Bennett AE, Jobe BA, Eisen GM, Fennerty MB, Hunter JG, Fleischer DE, Sharma VK, Hawes RH, Hoffman BJ, Rothstein RI, Gordon SR, Mashimo H, Chang KJ, Muthusamy VR, Edmundowicz SA, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Falk GW, Kimmey MB, Madanick RD, Chak A, Lightdale CJ. Radiofrequency ablation in Barrett's esophagus with dysplasia. N Engl J Med. 2009 May 28;360(22):2277-88. doi: 10.1056/NEJMoa0808145. PMID 19474425
- [Result] Shaheen NJ, Overholt BF, Sampliner RE, Wolfsen HC, Wang KK, Fleischer DE, Sharma VK, Eisen GM, Fennerty MB, Hunter JG, Bronner MP, Goldblum JR, Bennett AE, Mashimo H, Rothstein RI, Gordon SR, Edmundowicz SA, Madanick RD, Peery AF, Muthusamy VR, Chang KJ, Kimmey MB, Spechler SJ, Siddiqui AA, Souza RF, Infantolino A, Dumot JA, Falk GW, Galanko JA, Jobe BA, Hawes RH, Hoffman BJ, Sharma P, Chak A, Lightdale CJ. Durability of radiofrequency ablation in Barrett's esophagus with dysplasia. Gastroenterology. 2011 Aug;141(2):460-8. doi: 10.1053/j.gastro.2011.04.061. Epub 2011 May 6. PMID 21679712
- [Result] Phoa KN, van Vilsteren FG, Weusten BL, Bisschops R, Schoon EJ, Ragunath K, Fullarton G, Di Pietro M, Ravi N, Visser M, Offerhaus GJ, Seldenrijk CA, Meijer SL, ten Kate FJ, Tijssen JG, Bergman JJ. Radiofrequency ablation vs endoscopic surveillance for patients with Barrett esophagus and low-grade dysplasia: a randomized clinical trial. JAMA. 2014 Mar 26;311(12):1209-17. doi: 10.1001/jama.2014.2511. PMID 24668102
- [Result] Bergman JJ, Zhang YM, He S, Weusten B, Xue L, Fleischer DE, Lu N, Dawsey SM, Wang GQ. Outcomes from a prospective trial of endoscopic radiofrequency ablation of early squamous cell neoplasia of the esophagus. Gastrointest Endosc. 2011 Dec;74(6):1181-90. doi: 10.1016/j.gie.2011.05.024. Epub 2011 Aug 15. PMID 21839994
- [Result] van Vilsteren FG, Alvarez Herrero L, Pouw RE, ten Kate FJ, Visser M, Seldenrijk CA, van Berge Henegouwen MI, Weusten BL, Bergman JJ. Radiofrequency ablation for the endoscopic eradication of esophageal squamous high grade intraepithelial neoplasia and mucosal squamous cell carcinoma. Endoscopy. 2011 Apr;43(4):282-90. doi: 10.1055/s-0030-1256309. Epub 2011 Mar 31. PMID 21455869
- [Result] Wang WL, Chang IW, Chang CY, Lin JT, Mo LR, Wang HP, Lee CT. Circumferential balloon-based radiofrequency ablation for ultralong and extensive flat esophageal squamous neoplasia. Gastrointest Endosc. 2014 Dec;80(6):1185-9. doi: 10.1016/j.gie.2014.07.025. Epub 2014 Sep 23. No abstract available. PMID 25257127
- [Result] Wang WL, Chang IW, Chen CC, Chang CY, Mo LR, Lin JT, Wang HP, Lee CT. Radiofrequency Ablation Versus Endoscopic Submucosal Dissection in Treating Large Early Esophageal Squamous Cell Neoplasia. Medicine (Baltimore). 2015 Dec;94(49):e2240. doi: 10.1097/MD.0000000000002240. PMID 26656367
- [Result] He S, Bergman J, Zhang Y, Weusten B, Xue L, Qin X, Dou L, Liu Y, Fleischer D, Lu N, Dawsey SM, Wang GQ. Endoscopic radiofrequency ablation for early esophageal squamous cell neoplasia: report of safety and effectiveness from a large prospective trial. Endoscopy. 2015 May;47(5):398-408. doi: 10.1055/s-0034-1391285. Epub 2015 Feb 10. PMID 25668428
- [Derived] Wang WL, Tsai YN, Hsu MH, Lin JT, Wang HP, Lee CT. Endoscopic background mucosal resurfacing to prevent metachronous recurrence of superficial esophageal squamous cell cancer after curative endoscopic submucosal dissection: randomized pilot study with 5-year follow-up (with video). Gastrointest Endosc. 2025 Jun;101(6):1145-1154. doi: 10.1016/j.gie.2024.11.003. Epub 2024 Nov 8. PMID 39521094